CLINICAL TRIAL: NCT00243997
Title: Study of the Effects of the Becoming Parents Program on Couples Becoming Parents for the First Time
Brief Title: Evaluation of the Efficacy of the Becoming Parents Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Pamela Jordan/Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 96-2009-C14; R01NR004912 (NIH)
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Pregnancy
Keywords: parents; fathers; mothers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Subjects receiving the Becoming Parents Program
  Interventions: Behavioral: Becoming Parents Program
- 2 (Placebo Comparator): Subjects not receiving the Becoming Parents Program
  Interventions: Behavioral: Becoming Parents Program

INTERVENTIONS:
Behavioral: Becoming Parents Program — Couple focused educational program for couples adding a new baby to the family-21 hours of workshops during pregnancy with two three hour workshops after the baby is born.

SUMMARY:
The primary aim of this study is to test the effectiveness of the Becoming Parents Program--a couple focused educational program for couples having a first child--on individual and couple well being and the parent-infant relationship over the first three years of parenthood.

Other aims of this study are to evaluate the cost of implementing the Becoming Parents Program; to describe changes in individual and couple well-being over time, viewing the transition to parenthood from a developmental perspective using data from the control group; examine the various variables in the study over time from pregnancy through three years post-birth.

DETAILED DESCRIPTION:
The transition to parenthood is extremely difficult for both mothers and fathers, yet education and support during this major life transition emphasize getting through labor and birth, rather than preparing couples for the many changes accompanying parenthood. The classes of the Becoming Parents Program provide information and skills for taking care of the couple relationship, taking care of self, interacting with the baby, and the many ways becoming parents changes peoples' lives.

The purpose of this study is to evaluate the effects of the Becoming Parents Program classes on individual well being (measured by symptoms of depression and stress, perceived health, risk behaviors, health practices, health resource utilization), couple well-being (measured by marital satisfaction and stability), and the parent-infant relationship (measured by observation of the mother feeding the baby and the father teaching the baby) over the first three years of parenthood. Information is gathered by paper-and-pencil questionnaires during pregnancy, and at six months, one year, two years, and three years post-birth and by observation of parent-infant interaction at three months post-birth and videotaping and coding of couple interaction at six months post-birth.

Hypotheses are that couples who receive the Becoming Parents Program classes as compared to the couples who do not will:

1. have higher levels of marital satisfaction
2. have lower levels of depression
3. have less symptoms of stress
4. have higher levels of marital stability
5. communicate more effectively about a problem issue
6. have higher levels of health and well-being
7. score higher on observational evaluations of parent-infant interaction
8. report they are more satisfied with parenting, their partner's involvement in parenting their child, and with who does what in their family

ELIGIBILITY:
Inclusion Criteria:

* married couples
* expecting the birth of a first child
* not more than 30 weeks pregnant

Exclusion Criteria:

* consider their couple relationship in immediate danger or breaking up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2002-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Scores on a marital satisfaction scale at 6 months, 1 , 2 , 3 post-birth | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth

SECONDARY OUTCOMES:
Scores on a depression rating scale | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth
Scores on a symptoms of stress measure | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth
Whether or not subject couples are still married | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth
Coding of how effectively couples communicate about a problem issue in their relationship as observed from a videotape of the couples interacting at 6 months post-birth | 6 mos post-birth
Individual participant ratings of their own health, their partner's health, their baby's health | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth
Identification of health risk behaviors and health practices | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth
Health resource utilization | 6 mos, 1 yr, 2 yrs, 3 yrs post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Jordan, PhD, Principal Investigator — Dept of Family & Child Nursing, University of Washington